CLINICAL TRIAL: NCT03473392
Title: One-stage Exchange Arthroplasty for Chronic Prosthetic Joint Infections
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0237
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Exchange of Prosthetic Joint; Prosthetic Joint Infection; One-step Exchange
Keywords: pre-treatment; antibiotherapy; prosthetic joint infection; treatment failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The results found in the literature do not allow to define objectively the indications respective for a one-step or a two-step exchange of prosthetic joint. Some criteria could help to decide for one-step exchange or two-step exchange: bacteria is/are identified, profile of the bacteria, anesthetic difficulties,..

A puncture could allow to identify the bacteria involved in the prosthetic joint infection (PJI) and an antibiotherapy for a few days can be given to the patient in order to decrease the inoculum. Then, a one-step exchange can be performed.

The purpose of this study is to describe the management of patients who had a pre-treatment before a one-step exchange of their prosthetic joint.

ELIGIBILITY:
Inclusion Criteria:

* patient with prosthetic joint infection and having had a pre-treatment, managed at the Croix-Rousse Hospital
* > 18 years old

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having had puncture which allowed to identify bacteria responsible for the IPA and having had a pre-treatment for a few days against those bacteria before a one-step exchange of prosthetic joint
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
bacterial epidemiology | at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  This outcome will describe the bacterial epidemiology identified with a punction, the antibiotherapy used for pre-treatment, the characteristics of patients and the PJI.

SECONDARY OUTCOMES:
Treatment failure | at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

CONTACTS AND LOCATIONS:
Overall Officials: Tristan FERRY, Principal Investigator — Hospices Civils de Lyon